CLINICAL TRIAL: NCT06077786
Title: An Interventional Randomized, Double-blind, Placebo and Active Comparator-controlled, Four-way Crossover Trial Investigating the Analgesic Properties of a Single Oral Dose of Lu AG06474 in Healthy Participants
Brief Title: A Trial Investigating the Pain-relieving Properties of Lu AG06474 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20435A; 2023-503987-18-00 (Other: CTIS)
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Ibuprofen; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: Lu AG06474 + Placebo (Experimental): Participants will receive a single dose of Lu AG06474 (oral solution) and a single dose of placebo (3 placebo capsules).
  Interventions: Drug: Lu AG06474; Drug: Placebo
- Part B: Ibuprofen + Placebo to Lu AG06474 (Experimental): Participants will receive a single dose of ibuprofen (3 ibuprofen capsules) and a single dose of placebo to Lu AG06474 (oral solution).
  Interventions: Drug: Placebo to Lu AG06474; Drug: Ibuprofen
- Part C: Pregabalin + Placebo to Lu AG06474 (Experimental): Participants will receive a single dose of pregabalin (1 capsule + 2 placebo capsules) and a single dose of placebo to Lu AG06474 (oral solution).
  Interventions: Drug: Placebo to Lu AG06474; Drug: Pregabalin; Drug: Placebo
- Part D: Placebo to Lu AG06474 + Placebo (Experimental): Participants will receive a single dose of placebo to Lu AG06474 (oral solution) and a single dose of placebo (3 placebo capsules).
  Interventions: Drug: Placebo to Lu AG06474; Drug: Placebo

INTERVENTIONS:
Drug: Lu AG06474 — Oral solution
  Arms: Part A: Lu AG06474 + Placebo
Drug: Placebo to Lu AG06474 — Oral solution
  Arms: Part B: Ibuprofen + Placebo to Lu AG06474; Part C: Pregabalin + Placebo to Lu AG06474; Part D: Placebo to Lu AG06474 + Placebo
Drug: Ibuprofen — Capsule
  Arms: Part B: Ibuprofen + Placebo to Lu AG06474
Drug: Pregabalin — Capsule
  Arms: Part C: Pregabalin + Placebo to Lu AG06474
Drug: Placebo — Capsule
  Arms: Part A: Lu AG06474 + Placebo; Part C: Pregabalin + Placebo to Lu AG06474; Part D: Placebo to Lu AG06474 + Placebo

SUMMARY:
The main goal of this trial is to learn about the effect of Lu AG06474 on a battery of Evoked Pain Tests when a single dose is given to healthy adult participants. The effects of Lu AG06474 will be compared with 2 approved pain-relieving medications (ibuprofen and pregabalin) and with a placebo (a treatment that looks like the trial treatment but does not have any medicine in it). Each participant will receive 1 dose of each of these treatments during the trial (Lu AG06474, ibuprofen, pregabalin, and placebo), with 1 week between treatments. All treatments will be taken orally (by mouth), either as a liquid or a capsule.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) ≥18.5 and ≤32 kilograms per meter squared (kg/m^2) at the Screening Visit and at the Trial Baseline Visit.
* The participant is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, a neurological examination, vital signs, an ECG, and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The participant is a member of the site staff or of their immediate families or is a subordinate (or immediate family member of a subordinate) to any of the site staff.
* The participant has Fitzpatrick skin type IV, V and VI, wide-spread acne, tattoos, or scarring interfering with the area of interest (that is, upper back).
* The participant is currently enrolled in another clinical trial or used any investigational drug or device within 3 months (or <5 half-lives of that product, whichever is longer) prior to dose of investigational medicinal product (IMP), or has participated in more than 4 investigational drug studies within 1 year prior to Screening.
* The participant takes any disallowed medication within 14 days from first dose of trial drug.
* The participant has been vaccinated ≤14 days prior to the first dose of IMP.
* The participant is pregnant, breastfeeding, intends to become pregnant, or is of child bearing potential and not willing to use adequate contraceptive methods.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Pain Detection Thresholds (PDTs) for the UVB Heat Pain Test | Baseline to 6 hours post-dose
  The PDT is the degrees Celsius where the participant first detects pain.
Change From Baseline in Pain Detection Thresholds (PDTs) for the Capsaicin Heat Pain Test | Baseline to 6 hours post-dose
  The PDT is the degrees Celsius where the participant first detects pain.
Change From Baseline in Area of Secondary Mechanical Allodynia After the Capsaicin Challenge | Baseline to 6 hours post-dose
  The area of secondary mechanical allodynia will be reported for the capsaicin challenge, measured in squared millimeters (mm^2).
Change From Baseline in Pain Tolerance Thresholds (PTTs) for the Cold Pressor Test | Baseline to 6 hours post-dose
  The PTT is the timepoint (in seconds) where the participant can no longer tolerate the pain.
Change From Baseline in Pain Detection Thresholds (PDTs) for the Cold Pressor Test | Baseline to 6 hours post-dose
  The PDT is the timepoint (in seconds) where the participant first detects the pain.

SECONDARY OUTCOMES:
AUC0-8h: Area Under the Curve Concentration-time Curve from Zero to 8 hours Post-dose | 0 (predose) to 8 hours postdose on Day 1 to Day 22
Cmax: Maximum Observed Plasma Concentration | 0 (predose) to 8 hours postdose on Day 1 to Day 22
tmax: Nominal Time Corresponding to the Occurrence of Cmax | 0 (predose) to 8 hours postdose on Day 1 to Day 22
Difference to Placebo in Blood Levels of Endocannabinoids | 0 (predose) to 8 hours postdose on Day 1 to Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands